CLINICAL TRIAL: NCT06110247
Title: Evaluation of Renal Oxygenation in Pediatric Retrograde Intrarenal Surgery (RIRS) and Ureteroscopy (URS) Procedures by Near Infrared Spectroscopy (NIRS)
Brief Title: Evaluation of Renal Oxygenation by NIRS in Pediatric Endourologic Stone Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Şengül Özmert, Assoc. Prof. MD, Ankara City Hospital Bilkent
Other Study IDs: NIRS
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Renal Stone; Kidney; Complications; Ureter Stone; Renal Oxygenation
Keywords: Near infrared spectroscopy; Pediatric; Renal oxygenation; Endourologic stone surgery; infectious complication
MeSH Terms: conditions — Nephrolithiasis; Ureterolithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group R: Pre- and Postoperative hemoglobin (Hb), hematocrit (Htc), leukocyte (WBC), blood urea nitrogen (BUN), serum creatinine (sCr), procalcitonin, interleukin-6 and CRP values will be recorded. NIRS monitoring will be performed in addition to routine ASA monitoring. After the positions of the renal NIRS probes are confirmed by ultrasonography, the average value of the three measurements will be taken and the regional oxygen saturation index (rSO2) will be accepted as the initial value. NIRS, pulse oximetry, and hemodynamic data will be recorded every 5 minutes until recovery from anesthesia just prior to induction. When comparing the NIRS values measured during follow-up with the baseline NIRS value, a decrease of 20% or more than 20% will be considered significant. Anesthesia and surgery times will also be recorded. Postoperative fever and the amount of irrigation fluid used during the surgical procedure will be recorded .
  Interventions: Device: NIRS; Other: Taking a blood sample
- Group U: Pre- and Postoperative hemoglobin (Hb), hematocrit (Htc), leukocyte (WBC), blood urea nitrogen (BUN), serum creatinine (sCr), procalcitonin, interleukin-6 and CRP values will be recorded. NIRS monitoring will be performed in addition to routine ASA monitoring. After the positions of the renal NIRS probes are confirmed by ultrasonography, the average value of the three measurements will be taken and the regional oxygen saturation index (rSO2) will be accepted as the initial value. NIRS, pulse oximetry, and hemodynamic data will be recorded every 5 minutes until recovery from anesthesia just prior to induction. When comparing the NIRS values measured during follow-up with the baseline NIRS value, a decrease of 20% or more than 20% will be considered significant. Anesthesia and surgery times will also be recorded. Postoperative fever and the amount of irrigation fluid used during the surgical procedure will be recorded .
  Interventions: Device: NIRS; Other: Taking a blood sample
- Group H: The study involves continuous NIRS monitoring in addition to routine ASA monitoring. To establish the initial value of regional oxygen saturation (rSO2), renal NIRS probes will be positioned using ultrasonography, and an average of three measurements will be taken. Throughout the procedure, NIRS data, along with pulse oximetry and hemodynamic data, will be recorded at 5-minute intervals until the patient recovers from anesthesia just prior to induction. Significant changes in NIRS values will be determined if a decrease of 20% or more compared to the baseline measurement is observed. Anesthesia and surgery times will also be recorded.
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — After the positions of the renal NIRS probes are confirmed by ultrasonography, the average value of the three measurements will be taken and the regional oxygen saturation index (rSO2) will be accepted as the initial value.
Other: Taking a blood sample — Pre- and Postoperative hemoglobin (Hb), hematocrit (Htc), leukocyte (WBC), blood urea nitrogen (BUN), serum creatinine (sCr), procalcitonin, interleukin-6 and CRP values will be recorded.
  Groups: Group R; Group U

SUMMARY:
The study aims to compare renal oxygenation levels in retrograde intrarenal surgery (RIRS) and ureteroscopy (URS) procedures with a control group. Additionally, it seeks to determine if there is a connection between postoperative infection parameters and intraoperative renal oxygenation measurements.

DETAILED DESCRIPTION:
The study will involve ASA class I-III pediatric patients aged 1-18 undergoing RIRS, URS, and hypospadias surgery under general anesthesia. Patients will be divided into three groups: Group R (RIRS), Group U (URS), and Group H (Hypospadias/Control). Data collection will include patient height and weight. In Groups R and U, pre- and postoperative measurements such as hemoglobin, hematocrit, leukocyte count, BUN, serum creatinine, procalcitonin, interleukin-6, and CRP values will be recorded.

All three groups will undergo NIRS monitoring alongside routine ASA monitoring. Renal NIRS probes will be positioned using ultrasonography, and the average of three measurements will determine the regional oxygen saturation index (rSO2) as the initial value. NIRS, pulse oximetry, and hemodynamic data will be recorded every 5 minutes until recovery from anesthesia just prior to induction. A decrease of 20% or more than 20% when comparing NIRS values during follow-up with the baseline will be considered significant. The study will also document anesthesia and surgery times, as well as postoperative fever and the amount of irrigation fluid used in Groups R and U.

ELIGIBILITY:
Inclusion Criteria:

* 1-18 years ASA I-III class,
* Patients who will undergo RIRS, URS and Hypospadias surgeries under standard general anesthesia.
* Patients whose informed consent form is approved by their parents will be included in the study.

Exclusion Criteria:

* Exclusio criteria were the history of renal failure, renal tumors, infection of the perirenal region; receiving colloid or blood transfusion, having abscess, body mass index (BMI) not in the normal limits (≤3% or ≥97%)
* Patients whose parents do not approve the informed consent form will not be included in the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Due to the patient population of the hypospadias operation, Group H will consist of only male patients.
Study Population: ASA I-III class between the ages of 1-18, patients who will undergo RIRS and URS surgery under standard general anesthesia, as well as patients who will undergo hypospadias surgery (without a history of stones or kidney problems).
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Near infrared spectroscopy (NIRS) | NIRS values will be documented immediately prior to induction and every 5 minutes until recovery from anesthesia.
  Rretrograde intrarenal surgery (RIRS), ureteroscopy (URS) and hypospadias operations, renal oxygen level will be measured via NIRS monitor.

SECONDARY OUTCOMES:
Infection parameters | Preoperative and postoperative 24th hour
  Procalcitonin
Infection parameters | Preoperative and postoperative 24th hour
  Interleukin-6
Infection parameters | Preoperative and postoperative 24th hour
  C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital,Department Of Anesthesiology and Reanimation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No